CLINICAL TRIAL: NCT05536388
Title: Drug Discovery for Parkinson's With Mutations in the GBA Gene
Status: Recruiting | Type: Observational
Sponsor: New York Stem Cell Foundation Research Institute (Other)
Collaborators: Silverstein Foundation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 10-008
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-07

CONDITIONS: Parkinson Disease; Gaucher Disease; Healthy; GBA Gene Mutation
Keywords: Parkinson Disease; GBA Gene Mutation
MeSH Terms: conditions — Parkinson Disease; Gaucher Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsy (2-3mm) and/or blood (up to 50 mL); saliva; excess/leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Parkinson's Disease: Subjects in this group will have a diagnosis of Parkinson's disease with or without a known GBA gene mutation.
  Interventions: Other: Biological Sample Collection
- Gaucher Disease: Subjects in this group with have a diagnosis of Gaucher disease with or without a known GBA gene mutation.
  Interventions: Other: Biological Sample Collection
- Healthy Control: Subjects in this group will serve as healthy controls.
  Interventions: Other: Biological Sample Collection

INTERVENTIONS:
Other: Biological Sample Collection — Skin biopsy (2-3mm) and/or blood (up to 50 mL); saliva; excess/leftover biospecimens that were (or will be) collected for other purposes (e.g., medical procedure)
  Other Names: Biological sample collection for biobanking and research

SUMMARY:
The New York Stem Cell Foundation (NYSCF) Research Institute is performing this research to accelerate Parkinson's disease research and drug development by using cells from the body (such as skin or blood cells) to make stem cells and other types of cells, conduct research on the samples, perform genetic testing, and/or store the samples for future use.

Through this research, researchers hope to identify future treatments or even cures for Parkinson's disease.

DETAILED DESCRIPTION:
Researchers at the New York Stem Cell Foundation (NYSCF) Research Institute study diverse diseases, conditions, and traits by creating stem cells from biological samples. These "pluripotent" stem cells can become any cell in the human body, including cells that may be difficult, invasive, or impossible to obtain directly.

Additionally, researchers perform genetic testing to learn more about DNA, a material in most cells that contains instructions for the body's development and functions (such as traits like eye color and risk of certain diseases). A piece of DNA that determines the specific role of a cell is called a "gene." If the instructions in a gene are abnormal, this can lead to disease.

Participation in the study involves: (1) completion of health questionnaires, (2) providing a skin and/or blood sample from which stem cells may be created, (3) collection of a saliva sample for genetic analysis, and (4) possible future follow-up to provide additional information or learn about other research studies.

This study is not a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Diagnosis of Parkinson's disease, Gaucher disease, or healthy control.
* Must provide written informed consent unless physical limitations preclude signing.

Exclusion Criteria:

* For skin samples collected specifically for this study: history of keloid formation, coagulation disorder, allergy to the anesthetic, or anticoagulation use that precludes sample collection.
* For blood samples collected specifically for this study: coagulation disorder or other medical condition(s) that increases the risks associated with blood collection.
* For all prospective sample collections: Subjects who refuse to adhere to NYSCF's and/or a collection site's safety protocols will be excluded. Subjects with an AIDS diagnosis and CD4 count of less than 200 cells per microliter (mcL) of blood will be excluded due to increased risk of infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with a diagnosis of one or more of the listed conditions.
  Individuals without a condition to serve as healthy controls (a comparison group for those with conditions).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Establishment of a diverse bank of biological samples, stem cell lines, derivatives, and associated information. | Baseline
  Establish a robust disease signature using a cohort of PD and carefully matched control samples to screen a library of approximately 3,000 compounds to determine whether any compounds improve or reverse disease phenotypes.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Andres-Martin, Principal Investigator — New York Stem Cell Foundation Research Institute
Locations (1):
- The New York Stem Cell Foundation Research Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No